CLINICAL TRIAL: NCT04957095
Title: Motor Network Physiology Characterization During Deep Brain Stimulation Surgery
Brief Title: Motor Network Physiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nader Pouratian, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2021-0376; 1R01NS097782-01A1 (NIH)
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Essential Tremor
Keywords: deep brain stimulation; levodopa medication; motor cortex; basal ganglia; thalamus
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: Basic science study of effects of therapeutic interventions on intracranial physiology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's disease patients (Experimental): This group consists of Parkinson's disease patients who are undergoing deep brain stimulation surgery for treatment of their movement disorder. Participants will complete behavioral assessments while receiving subcortical DBS stimulation and / or inhaled levodopa medication, Inbrija. Stimulation will be applied at the previously determined therapeutic frequency. Two capsules (84 mg) of Inbrija will be administered.
  Interventions: Drug: Apomorphine Injectable Solution; Other: Subcortical Stimulation

INTERVENTIONS:
Drug: Apomorphine Injectable Solution — Apomorphine injected for therapeutic relief
Other: Subcortical Stimulation — Subcortical simulation of the deep brain stimulation surgery target site will be applied by clinically placed deep brain stimulation electrodes at the previously determined therapeutic setting

SUMMARY:
The brain networks controlling movement are complex, involving multiple areas of the brain. Some neurological disorders, like Parkinson's disease (PD) and essential tremor (ET), cause abnormalities in these brain networks. Deep brain stimulation is a treatment that is used to treat these types of neurological diseases and is thought to help patients by modulating brain networks responsible for movement. Levodopa medication is also used to modulate this brain networks in patients with PD. The overall objective is to develop a unified theory of basal ganglia thalamocortical (BGTC) circuit dynamics that accounts for disease symptomatology, movement, and their inter-relationship. The underlying hypothesis, is that the rigidity and bradykinesia of PD are fundamentally related to excessive functional coupling across nodes in the BGTC motor circuit impeding effective information flow. In this research, the investigator will take advantage of the unique opportunity provided by awake deep brain stimulation surgery to learn more about how the brain functions in a diseased state and how deep brain stimulation changes these networks to make movement more normal. The investigator will simultaneously assess cortical and subcortical electrophysiology in relation to clinical symptoms and behavioral measures and in response to deep brain stimulation, cortical stimulation, and pharmacologic therapy in patients undergoing Deep Brain Stimulation (DBS) implantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease who have been recommended to undergo deep brain stimulation for management of their movement disorder
* Preoperative MRI without evidence of cortical or subdural adhesions or vascular abnormalities
* Willingness and ability to cooperate during conscious operative procedure for up to 40 minutes

Exclusion Criteria:

* Patients with recent use (within one week) of anticoagulant or antiplatelet agents
* Neurocognitive testing indicating amnestic cognitive deficits

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
cortical ECoG and subcortical recordings | baseline
  Cortical ECoG and subcortical LFP recordings will occur during DBS implantation surgery during the behavioral assessments and/or Inbrija administration.
Behavioral assessment | baseline
  Each patient will complete a task that assesses the kinematics of movement, self-initiation of movement, and/or effect of Inbrija on movement

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No